CLINICAL TRIAL: NCT00461084
Title: Biaxin(Clarithromycin)Based Antibiotic Therapy In Previously Untreated, Advanced Stage Indolent Lymphoma
Brief Title: Biaxin Based Antibiotic Therapy in Previously Untreated, Advanced Stage Indolent Lymphoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-038
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Lymphoma
Keywords: Lymphoma; Advanced Stage; Untreated; Advanced Stage Lymphoma; Untreated Lymphoma; 07-038
MeSH Terms: conditions — Lymphoma | interventions — Clarithromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue and whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: lymphoma follicular
  Interventions: Drug: BIAXIN (CLARITHROMYCIN)
- 2: lymphoma non-follicular
  Interventions: Drug: Biaxin (clarithromycin)

INTERVENTIONS:
Drug: BIAXIN (CLARITHROMYCIN) — Biaxin (clarithromycin) 500 mg will be administered by mouth twice daily for 12 weeks in all patients. In H. pylori positive patients, Prevpak standard therapy (lansoprazole, amoxicillin, clarithromycin) will be administered for the first 2 weeks.Following Biaxin (clarithromycin) antibiotic therapy, the patient will be reassessed for eradication of H. pylori if previously present.
  Groups: 1
Drug: Biaxin (clarithromycin) — Biaxin (clarithromycin) 500 mg will be administered by mouth twice daily for 12 weeks in all patients. In H. pylori positive patients, Prevpak standard therapy (lansoprazole, amoxicillin, clarithromycin) will be administered for the first 2 weeks.Following Biaxin (clarithromycin) antibiotic therapy, the patient will be reassessed for eradication of H. pylori if previously present.
  Groups: 2

SUMMARY:
The purpose of this study is to see if a treatment with Biaxin (clarithromycin) which is an antibiotic given by mouth for 3 months can delay the growth of your lymphoma or shrink the lymphoma. We would also like to see how Biaxin (clarithromycin) works on lymphoma and blood cells.There is some evidence that this medication may change the behavior of lymphocytes, in addition to its known anti-infection activity.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate a biaxin (clarithromycin)-based antibiotic therapy in previously untreated patients with indolent lymphoma who do not require active lymphoma therapy (utilizing GELF criteria,). This is the primary objective Response rate (CR + PR) stratified for Follicular/Non-Follicular disease.

The secondary objectives of this study are to understand the biologic correlates of indolent lymphoma biaxin (clarithromycin) response and progression:

Response rate (CR + PR) according to H. pylori positive or negative (RR with a confidence interval will be estimated for each subset). Immunohistochemistry in all diagnostic biopsy specimens: Lymphocyte- Activated Macrophage (CD68) and other selected markers to clarify tumor infiltrating cells. Peripheral blood mononuclear cell (PBMCs) studies to evaluate possible HDAC (histone deacetylase) inhibition with biaxin (clarithromycin) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of follicular lymphoma: grades I, II, or IIIA, or non-follicular lymphoma: lymphoplasmacytoid lymphoma, small lymphocytic lymphoma, marginal B-cell lymphoma, or MALT lymphoma (as defined in the WHO classification1) as reviewed by a hematopathologist at Memorial Hospital.
* Staging fulfills criteria for no initial treatment according to GELF criteria for advanced stage disease. None of the following should be present:

  * A nodal or extranodal mass with a diameter of >7 cm,
  * Involvement of at least three nodal sites [each with a diameter of >3 cm],
  * Systemic symptoms,
  * Symptomatic splenomegaly,
  * Ureteral compression.
  * No prior treatment for lymphoma is permitted.
  * Measurable disease is required.
  * Karnofsky performance status > 70%
  * The patient may not have a previous history of radiation therapy.
  * Patient or guardian must be able to sign voluntary written consent.
  * Male or female patients 18 years of age or greater.

Exclusion Criteria:

* Allergy to biaxin (clarithromycin), erythromycin, or other macrolide antibiotic. Patients requiring use of ergot derivatives, pimozide, cisapride, or astemizole; combination with ranitidine bismuth citrate should not be used in patients with history of acute porphyria or CrCl <25 mL/minute.
* Prior treatment with Biaxin (clarithromycin) during the prior 6 months.
* Histologic diagnosis of follicular grade 3B or aggressive non-Hodgkin's lymphoma.
* Histologic evidence of transformation from low grade/indolent NHL to aggressive NHL.
* Prior treatment for non-Hodgkin's lymphoma.
* Regional lymphoma (peripheral stages I and II) eligible for involved field irradiation.
* GELF criteria21 for institution of systemic chemotherapy, which includes:

  * A nodal or extranodal mass with a diameter of >7 cm,
  * Involvement of at least three nodal sites [each with a diameter of >3 cm],
  * Systemic symptoms,
  * Symptomatic splenomegaly,
  * Ureteral compression.
* Patients with a known history of HIV, Hepatitis B or C seropositivity.
* Patients who require therapy with systemic corticosteroids.
* Prior history of malignancy within the past five years or a concurrent malignancy, with the exceptions of cutaneous basal cell carcinoma or carcinoma in situ of the uterine cervix.
* Pregnant or lactating women, since imaging cannot be done in this setting.18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously Untreated follicular lymphoma or non-follicular lymphoma will be recrited at MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate a biaxin (clarithromycin)-based antibiotic therapy in previously untreated patients with indolent lymphoma who do not require active lymphoma therapy (utilizing GELF criteria,). | conclusion of study

SECONDARY OUTCOMES:
The secondary objectives of this study are to understand the biologic correlates of indolent lymphoma biaxin (clarithromycin) response and progression | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Carol Portlock, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Portlock CS, Hamlin PA, Gerecitano JF, Noy A, Palomba ML, Walkley J, Corcoran S, Migliacci J, Schoder H, Papanicolaou G, Markowitz AJ. A Positive Prospective Trial of Antibiotic Therapy in Advanced Stage, Non-Bulky Indolent Lymphoma. Tumor Microenviron Ther. 2015 Feb;2(1):14-18. doi: 10.1515/tumor-2015-0001. Epub 2015 Feb 18. PMID 26798624
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org